CLINICAL TRIAL: NCT05162404
Title: Patient-Centered Video Education Intervention to Improve Rural Cancer Care Delivery
Brief Title: Video Education to Improve Rural Cancer Care Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: The Hope Foundation for Cancer Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Okado 2021-1
Record Dates: First submitted 2021-10-27; First posted 2021-12-17 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video Intervention (Experimental): The intervention in this study is a TED-talk style video series designed to provide patient education on cancer, care coordination, and self-advocacy. The content is designed to provide both a background about cancer disease and to address each of the specific domains in care coordination (CCI). The development of video contents was informed by our prior/current research in rural care coordination and components of evidence-based interventions including the patient navigator training by the George Washington University Cancer Institute, Imi Hale (the Native Hawaiian Cancer Network), and a supportive care intervention by Mokuau et al. As the target population of this intervention is rural patients, videos include some rural-specific considerations related to care coordination.
  Interventions: Behavioral: Video Education Program

INTERVENTIONS:
Behavioral: Video Education Program — The following topics are addressed in each module of the videos:
  1. Understanding cancer and cancer treatment - including an understanding of stage, site of origin, metastases, treatment options, toxicities and anticipated outcomes.
  2. Care coordination basics (CC: Communication) - including navigating care related to appointments, how to handle issues after-hours, and the expected roles of other healthcare providers (e.g., PCPs).
  3. How to be a self-advocate (CC: Navigation and Operational) - including how to ask questions, being empowered to talk to your doctor, when a second opinion is needed, when to explore clinical trials, and how to best incorporate a caregiver into your treatment.

SUMMARY:
The purpose of this study is to understand if a video-based education program delivered on a tablet device will improve care coordination experiences for patients with cancer living in rural areas.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a newly diagnosed Stage I, II, or III disease at the time of enrollment.
* Patients to be treated with adjuvant chemotherapy or recent initiation of (within 1 month of starting) adjuvant chemotherapy.
* Patients with a history of previous malignancy treated with chemotherapy within the last 3 years are not eligible, as their perceptions of care coordination may be impacted by their previous treatment.
* Patients must be ≥ 18 years of age.
* Patients must be able to read, write, and speak English. Study materials and telephone calls are only available in English.
* Patients must be residents of Hawaii, Kauai, or Maui counties
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in rural patients' perceptions of cancer care coordination as assessed by the Care Coordination Instrument at 4-6 months post-intervention. | 6 months

SECONDARY OUTCOMES:
Rural patient satisfaction with video education materials as assessed by semi-structured telephone interview. | 6 months
To examine patient demographic and clinical information collected from the background questionnaire as potential correlates of patients' perceptions of cancer care coordination at post-intervention | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hawaii Cancer Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okado I, Braun-Inglis C, Matsumoto K, Elhajj C, Cassel K, Berenberg J, Holcombe RF. Feasibility of a Remote Patient Video Education Intervention to Improve Care Coordination for Rural Cancer Patients. J Cancer Educ. 2025 Aug;40(4):594-599. doi: 10.1007/s13187-024-02550-6. Epub 2024 Dec 5. PMID 39636502